CLINICAL TRIAL: NCT02916199
Title: Primary Needle Knife Fistulotomy Versus Conventional Cannulation Method in Patients With High Risk of Post-endoscopic Retrograde Cholangiopancreatography Pancreatitis: A Multicenter Randomized Controlled Trial
Brief Title: Primary Needle Knife Fistulotomy Versus Conventional Cannulation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung III Jang, Assistant professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2017-0092
Record Dates: First submitted 2016-09-24; First posted 2016-09-27 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Common Bile Duct Stone; Malignant Hepatobiliary Neoplasm; Biliary Stricture; Pancreatic Diseases; Sphincter of Oddi Dysfunction
MeSH Terms: conditions — Gallstones; Pancreatic Diseases; Sphincter of Oddi Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Needle knife fistulotomy (Experimental): Device: Needle knife fistulotomy Disease: Common bile duct stone, Malignant biliary stricture, Benign biliary stricture, Benign pancreatic disease, biliary sphincter of Oddi dysfunction Indication: High risk of post-endoscopic retrograde cholangiopancreatography pancreatitis
  - Intervention: canulation of ampulla of Vater Intervention: canulation of ampulla of Vater
  Interventions: Device: cannulation of ampulla of Vater
- conventional cannulation (Active Comparator): Device: conventional canulation catheter Disease: Common bile duct stone, Malignant biliary stricture, Benign biliary stricture, Benign pancreatic disease, biliary sphincter of Oddi dysfunction Indication: High risk of post-endoscopic retrograde cholangiopancreatography pancreatitis
  - Intervention: canulation of ampulla of Vater Intervention: canulation of ampulla of Vater
  Interventions: Device: cannulation of ampulla of Vater

INTERVENTIONS:
Device: cannulation of ampulla of Vater — Cannulation of ampulla of Vater is a procedure that a guide-wire is passed through ampulla using interventional devices

SUMMARY:
The aim of this study are to evaluate the feasibility of needle knife fistulotomy (NKF) as an initial procedure for biliary access in patients with biliary disease who are at increased risk for post-endoscopic retrograde endoscopic retrograde cholangiopancreatography (PEP) and to assess the incidence rate of complications including PEP between NKF and conventional cannulation methods.

DETAILED DESCRIPTION:
Endoscopic retrograde endoscopic retrograde cholangiopancreatography (ERCP) is widely used for the diagnosis and treatment of pancreatic and biliary tract disease. However, post-ERCP pancreatitis (PEP) is the most common adverse event following the procedure, ranging from 2% to 10% in nonselective cases, and it can cause substantial morbidity, mortality, or high medical costs. Recent advances in cannulation technique and accessories for biliary cannulation have contributed to reduce the incidence of PEP, but biliary cannulation can fail in 5% to 20% of cases of ERCP. Suprapapillary needle-knife fistulotomy (NKF), with or without large-diameter balloon dilation, has been used as a rescue method in cases of difficult biliary cannulation, and NKF was recommended as an initial approach to selective biliary cannulation in cases of repetitive unintentional pancreatic cannulation.9 Moreover, difficult biliary cannulation is known to be a risk factor for PEP, and it has been reported that NKF is associated with a low risk of PEP. Thus, we hypothesized that NKF may reduce the risk of PEP in patients who are at increased risk for PEP.

ELIGIBILITY:
Inclusion Criteria:

* Patient who submitted a written informed consent for the this trial, and 18 ~ 90 years old
* Patient who have naïve ampulla (no previous procedure was performed at ampulla)
* Patient who is suspected to have biliary obstruction or biliary disease
* Patient who is needed to have endoscopic retrograde cholangiopancreatography for treatment of biliary obstruction
* Patient who have risks of post-endoscopic retrograde cholangiopancreatography pancreatitis among bellows (at least one more);

  1. suspected biliary sphincter of Oddi dysfunction
  2. young age (18~50 years)
  3. female
  4. normal common bile duct diameter (≤9mm)
  5. normal serum bilirubin level
  6. Obesity (body mass index > 30)
  7. Past history of acute pancreatitis

Exclusion Criteria:

* Patient who is below 18 year old
* Patient who is pregnant
* Patient with mental retardation
* Patient is sensitive to contrast agents
* Patient who received sphincterotomy or pancreatobiliary operation previously
* Patient who have ampulla of Vater cancer
* Patient who have difficulty for approach to ampulla due to abdominal surgery including stomach cancer with Billroth II anastomosis
* Patient who have pancreatic diseases as bellow (at least one more);

  1. Patient who have acute pancreatitis within 30days before enrollment
  2. Patient who have idiopathic acute recurrent pancreatitis
  3. Patient who have pancreatic divisum
  4. Patient who have obstructive chronic pancreatitis
  5. Patient who pancreatic cancer
* Patients who have improper ampulla shape as bellows;

  1. Small ampulla (ampulla without oral protrusion)
  2. Flat or crooked or asymmetric ampulla
  3. Ampulla with peri-ampullary diverticulum type I or II

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence rate of post-endoscopic retrograde cholangiopancreatography | 1 week

SECONDARY OUTCOMES:
Incidence rate of complications including bleeding, perforation and infection | 1 week
Success rate of cannulation | 1 day
Success rate of stone removal | 1 day

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - CHA Bundang Medical Center, Seongnam, Bundang-gu
  - Gangnam Severance Hospital, Seoul, Gangnam-gu
  - Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do
  - In Ha University Hospital, Incheon, Jung-gu
  - Soon Chun Hyang University Hospital, Cheonan, Cheonan, Namdong-gu
  - Gachon University Gil Medical Center, Incheon, Namdong-gu
  - Pusan National University Hospital, Busan, Seo-gu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jang SI, Kim DU, Cho JH, Jeong S, Park JS, Lee DH, Kwon CI, Koh DH, Park SW, Lee TH, Lee HS. Primary Needle-Knife Fistulotomy Versus Conventional Cannulation Method in a High-Risk Cohort of Post-Endoscopic Retrograde Cholangiopancreatography Pancreatitis. Am J Gastroenterol. 2020 Apr;115(4):616-624. doi: 10.14309/ajg.0000000000000480. PMID 31913191